CLINICAL TRIAL: NCT05995210
Title: Comparing the Effectiveness of Kinesio Taping and Knee Orthosis in Patients with Patellofemoral Pain Syndrome: a Randomized Controlled Study
Brief Title: Comparing the Effectiveness of Kinesio Taping and Knee Orthosis in Patients with Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Yunus Özdemir, PhD, Physiotherapist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulMUH-DPTR-Yozdemir-0859
Record Dates: First submitted 2023-07-03; First posted 2023-08-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome; Patellofemoral Pain; Patellofemoral Syndrome; Orthotic Devices; Kinesiotape
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled single-blind
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Kinesio taping group (Experimental): In addition to the standard exercise program, kinesio taping was applied to the knee for 6 weeks.
  Interventions: Procedure: Kinesio taping; Procedure: Control
- Orthosis group (Experimental): In addition to the standard exercise program, they were asked to use a knee orthosis for 6 weeks.
  Interventions: Procedure: Orthosis; Procedure: Control
- Control group (Active Comparator): A standard exercise program was applied for 6 weeks.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Kinesio taping — A corrective kinesio taping was applied to the patellofemoral joint for the knee. In addition, exercise therapy was taken.
  Arms: Kinesio taping group
Procedure: Orthosis — They were asked to use a knee orthosis for a minimum of 6 hours a day. They also received exercise therapy.
  Arms: Orthosis group
Procedure: Control — An exercise program focused on the knee and hip muscles was given two days a week.

SUMMARY:
The aim of the study is to compare the efficacy of kinesio taping treatment and knee orthosis treatment in Patellofemoral Pain Syndrome (PFAS). 54 patients were included in the study and the patients were divided into 3 groups as kinesio taping group (KTG) (n=18), orthotics group (OG) (n=18) and control group (CG) (n=18). A progressive exercise program was applied to all groups and patients were treated 2 days a week for 6 weeks.While kinesio taping was applied to KTG in each session, knee orthosis was given to OG and they were asked to use it for 6 weeks. Visual Analogue Scale (VAS), Kujala Score, Knee injury and Osteoarthritis Outcome Score (KOOS) and isokinetic strength test (IST) were used in the evaluation.

DETAILED DESCRIPTION:
Patients were divided into 3 groups as patellofemoral knee orthosis group, kinesio taping group and control group. Randomization of group allocation was done using the website "https://www.randomizer.org". Patients were unaware of the other group's treatment program and group allocation. All participants signed an informed consent form before the study. The primary outcome measure of our study was the Kujala Score, and the secondary outcome measures were the Knee Injury and Osteoarthritis Outcome Score (KOOS), Visual Analog Scale (VAS), quadriceps and hamstring isokinetic muscle strength. The evaluations were performed before and after treatment. All patients were informed about the disease and treatment process before treatment. Patients were informed about the things they should pay attention to for pain management in daily life activities and suggestions were made. In addition, all patients received at least 2 weeks of NSAID treatment by the orthopedist. A progressive exercise program was applied to all treatment groups. The progressive exercise program was continued under the supervision of a physiotherapist 2 days a week for 6 weeks. The progressive exercise program consisted of strengthening exercises for the muscles around the knee and hip, stretching exercises for the hamstring and gastrosoleus muscles. The knee orthosis group received the OrthoCare® 6158 Genucare Luxa knee orthosis. T-max Kinesiology Tape® (Tmax Medical Co., South Korea) brand kinesio tape was used in all patients. In kinesio tape application, 2 Y-shaped tapes were used. The activation technique was applied to the VMO muscle with the first band. In the second band, mechanical correction technique was applied to the patella.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-45
* Patients with a body mass index (BMI) less than 29.9
* Anterior knee pain defined as 3 points on the 10 cm Visual Analogue Scale when performing at least two activities of sitting for a long time, climbing/descending stairs, squatting, running and jumping

Exclusion Criteria:

* Patients with knee osteoarthritis
* History of surgery involving the lower extremity
* Patellar or quadriceps tendinopathy
* Injury to the meniscus or knee ligaments
* Patients showing an allergic response to kinesio tape
* Patients previously treated with PFAS
* Existing hip pathologies
* History of patellar subluxation or dislocation
* Patients with neurological disorders
* Patients who did not fill out the voluntary consent form

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Change in baseline Kujala scores of patients treated at week 6 | 6 weeks
  It is a score that evaluates symptoms and function in patients with patellofemoral pain syndrome. Patients were asked to complete this score before starting the treatment and again at the end of the 6-week treatment.

SECONDARY OUTCOMES:
Change in baseline Visual Analogue Scale of patients treated at week 6 | 6 weeks
  It is a scale that evaluates pain. Patients were asked to complete this scale before starting the treatment and again at the end of the 6-week treatment.
Change in baseline Knee Injury and Osteoarthritis Outcome Score of patients treated at week 6 | 6 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) is a score used to evaluate symptoms and functional status related to knee injury and knee osteoarthritis. Patients were asked to complete this score before starting the treatment and again at the end of the 6-week treatment.
Change in baseline isokinetic strength test of patients treated at week 6 | 6 weeks
  This test is a strength test performed with an isokinetic strength testing machine. This test was applied to the patients before starting the treatment and at the end of the 6-week treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Özdemir, MSc, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No